CLINICAL TRIAL: NCT02051387
Title: Cannabidiol as a Different Type of an Antipsychotic: Drug Delivery and Interaction Study With Approved Antipsychotics in Vivo
Brief Title: Cannabidiol as a Different Type of an Antipsychotic: Drug Delivery and Interaction Study
Acronym: CBD-IS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-IS; 2008-008245-38 (EudraCT Number)
Record Dates: First submitted 2013-09-18; First posted 2014-01-31 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol; Amisulpride; Olanzapine; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cannabidiol (Active Comparator): Cannabidiol capsule, 200 mg single dose
  Interventions: Drug: Cannabidiol
- Cannabidiol CR (Experimental): Cannabidiol tablet, various dosages
  Interventions: Drug: Cannabidiol CR
- Amisulpride and Cannabidiol CR (Experimental): Interaction between Amisulpride and Cannabidiol CR
  Interventions: Drug: Cannabidiol CR; Drug: Amisulpride
- Olanzapine and Cannabidiol CR (Experimental): Interaction between Olanzapine and Cannabidiol CR
  Interventions: Drug: Cannabidiol CR; Drug: Olanzapine
- Quetiapine and Cannabidiol CR (Experimental): Interaction between Quetiapine and Cannabidiol CR
  Interventions: Drug: Cannabidiol CR; Drug: Quetiapine
- Risperidone and Cannabidiol CR (Experimental): Interaction between Risperidone and Cannabidiol CR
  Interventions: Drug: Cannabidiol CR; Drug: Risperidone
- Cannabidiol CR and Placebo (Placebo Comparator): Cannabidiol CR levels without interaction with antipsychotics
  Interventions: Drug: Cannabidiol CR; Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol CR
  Other Names: Arvisol
  Arms: Amisulpride and Cannabidiol CR; Cannabidiol CR; Cannabidiol CR and Placebo; Olanzapine and Cannabidiol CR; Quetiapine and Cannabidiol CR; Risperidone and Cannabidiol CR
Drug: Cannabidiol
  Arms: Cannabidiol
Drug: Amisulpride
  Arms: Amisulpride and Cannabidiol CR
Drug: Olanzapine
  Arms: Olanzapine and Cannabidiol CR
Drug: Quetiapine
  Arms: Quetiapine and Cannabidiol CR
Drug: Risperidone
  Arms: Risperidone and Cannabidiol CR
Drug: Placebo
  Arms: Cannabidiol CR and Placebo

SUMMARY:
Despite recent advances in the understanding and treatment of schizophrenia, this devastating disease still affects one percent of world's population. Existing antipsychotics reduce psychotic symptoms but are generally not very effective in treating so called negative symptoms such as blunted affect and social withdrawal or cognitive disturbances due to the disease. Furthermore, a significant portion of patients is refractory to all current treatments. Therefore new treatment strategies are needed.

Several studies suggest a strong association between schizophrenia and the endocannabinoid system. This system mediates e.g. the pro-psychotic effects of the best-known ingredient of the cannabis plant - delta-tetrahydrocannabinol (Δ9-THC). While the pro-psychotic Δ9-THC is known to abet the onset of schizophrenia, another, non-psychotomimetic plant ingredient - cannabidiol - has recently been shown to exert antipsychotic effects similar to those of one of the most effective modern antipsychotics, amisulpride, but it induced significantly less side effects.

In this phase I safety study, the investigators will evaluate the pharmacokinetics, pharmacoequivalence, and drug-drug interaction profile with current antipsychotics of a new tablet pharmaceutical preparation of cannabidiol in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* Both, female and male subjects may participate
* Age between 18 and 45
* Negative drug screening at the time of screening
* Non-smoking
* In female participants in fertile age, reliable contraception, which means contraception's pearl-index is equal or smaller than 1.
* Body Mass Index between 18 and 30

Exclusion Criteria:

* Lack of accountability
* Any current psychiatric disorder through the Structured Clinical Interview for DSM-IV (SCID) at the time of screening
* Pregnancy or lactation phase in female at the time of screening
* Any known psychiatric or neurological illness in the participant's history.
* Known family history concerning psychiatric disorders
* Relevant use of cannabis (which is defined on the present state of knowledge as at the most five times lifetime-consumption and no consumption for at least one year)
* Severe physical (internal) or neurological illness, especially cardiovascular, renal, advanced respiratory, haematological or endocrinological failures or infectious diseases (acute hepatitis A, B or C or HIV) assessed at the time of the screening by the subject's history, clinical examination and laboratory testing, at the discretion of the investigator
* Consumption of any illicit drugs (except cannabis in history, see above)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Plasma levels of cannabidiol | up to 10 days

SECONDARY OUTCOMES:
Area Under Curve (AUC) | up to 10 days
serum antipsychotic concentration | baseline and after seven days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Central Institute of Mental Health, Mannheim, Baden-Wurttemberg
  - Dept. of Pharmacology, University of Cologne, Cologne, North Rhine-Westphalia